CLINICAL TRIAL: NCT06111170
Title: Effect of Compression Dressing After Upper Eyelid Blepharoplasty on Edema, Ecchymosis, Pain and Ocular Surface Irritation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augenklinik LMU (Other)
Responsible Party: Principal Investigator, Anna Schuh, Dr. med. Anna Schuh, Consultant in Oculoplastics, FEBO, Augenklinik LMU
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-305
Record Dates: First submitted 2023-10-25; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Dermatochalasis of Eyelid

STUDY DESIGN:
Intervention Model Description: two arms. After randomization one eyelid of each patient was applied with a compression dressing, the other eyelid not.
Who Masked: Investigator
Masking Description: There was one blinded observer evaluating the results using pre and postoperative photographs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression dressing (Active Comparator): Compression dressing was applied to one of the eyelids which was chosen by randomization postoperatively
  Interventions: Device: Compression dressing
- no dressing (No Intervention): No dressing was applied on the other eyelid (control group)

INTERVENTIONS:
Device: Compression dressing — Application of dressing
  Arms: Compression dressing

SUMMARY:
Study to analyze whether there is a difference in postoperative outcome regarding edema, ecchymosis, pain, OSI and discomfort of the patients after blepharoplasty if a compression dressing is used or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper eyelid dermatochalasis who were scheduled for upper eyelid blepharoplasty

Exclusion Criteria:

* previous surgery on the upper eyelid, previous eye lid trauma, congenital lid changes, blepharochalasis syndrome, coagulation disorders or indication for combined ptosis and blepharoplasty surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Edema | Measures are taken the first day after surgery (D1), one week after surgery (D7) and eight weeks after surgery (D56)
  Degree of edema postoperatively, rated on a four point rating scale: 0 = no, 1 = minimal, 2 = moderate, 3 = severe

CONTACTS AND LOCATIONS:
Locations (1):
- Augenklink LMU, München, Germany

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from the corresponding author, [A.S.], upon reasonable request

REFERENCES:
- [Derived] Schuh A, Reischmann L, Hintschich CR. Effect of Compression Dressing After Upper Eyelid Blepharoplasty on Edema, Ecchymosis, Pain, and Ocular Surface Irritation. Ophthalmic Plast Reconstr Surg. 2024 Nov-Dec 01;40(6):627-633. doi: 10.1097/IOP.0000000000002666. Epub 2024 Apr 11. PMID 38624150